CLINICAL TRIAL: NCT01240681
Title: A Pilot Study of Blood Oxygen Level Dependent Magnetic Resonance Imaging (BOLD MRI) and Fluorothymidine Positron Emission Tomography (FLT PET) in Patients With Locally Advanced Breast Cancer Undergoing Neoadjuvant Chemotherapy
Brief Title: Blood Oxygen Level Dependent Magnetic Resonance Imaging (BOLD MRI) and Fluorothymidine Positron Emission Tomography (FLT PET) in Patients With Locally Advanced Breast Cancer Undergoing Neoadjuvant Chemotherapy
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCOG-2010-IMPACT
Record Dates: First submitted 2010-11-01; First posted 2010-11-15 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Locally Advanced Breast Cancer (LABC)
Keywords: Locally Advanced Breast Cancer (LABC); neoadjuvant chemotherapy; Fluorothymidine Positron Emission Tomography (FLT PET); Blood Oxygen Level Dependent Magnetic Resonance Imaging (BOLD MRI); tumor response; mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLT PET and BOLD MRI scan (Other): All subjects will have the study intervention of FLT PET and BOLD MRI at baseline and after the first cycle of chemotherapy
  Interventions: Procedure: FLT PET and BOLD MRI scan

INTERVENTIONS:
Procedure: FLT PET and BOLD MRI scan — Eligible consenting patients with LABC receiving neoadjuvant chemotherapy (NA CT) will undergo FLT PET, BOLD MRI, and clinical examination of the involved breast including ipsilateral axillary and supraclavicular nodes to assess the treatment response to chemotherapy (CT). The imaging studies will be performed at baseline and after the first cycle of NA CT.

SUMMARY:
The objective of this pilot study is to determine the effectiveness of Fluorothymidine Positron Emission Tomography (FLT PET) and Blood Oxygen Level Dependent Magnetic Resonance Imaging (BOLD MRI) in assessing tumour response to neoadjuvant chemotherapy (NA CT) in women with locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of breast cancer (invasive ductal or lobular carcinoma). Breast sarcoma and lymphoma are not eligible.
* Clinical diagnosis of locally advanced breast cancer (Stage IIB (T3,N0,M0), Stage IIIA, IIIB, or IIIC, according to American Joint Committee on Cancer (AJCC) Tumour-Node-Metastasis (TNM) Cancer Staging), including inflammatory breast cancer.
* Ability to undergo neoadjuvant chemotherapy.

Exclusion Criteria:

* Evidence of metastatic disease (identified on chest x-ray, liver ultrasound, bone scan or other imaging tests);
* Previous chemotherapy or hormonal therapy for breast cancer;
* Significant concurrent medical problems that result in the patient being unfit for surgery (e.g. uncontrolled diabetes, active cardiac disease, severe chronic obstructive pulmonary disease);
* Known pregnancy or lactating female (e.g. positive serum beta human chorionic gonadotropin (B-hCG) pregnancy test);
* Inability to lie supine for imaging with Positron Emission Tomography (PET);
* Any contraindication to undergoing Magnetic Resonance Imaging (MRI) or PET;
* Currently receiving Antabuse;
* Inability to provide informed consent (e.g. dementia or severe cognitive impairment).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Clinical response (partial and complete) | 6 months (approximately)
  Partial clinical response refers to at least a 50% reduction in the dimensions of the tumour mass and a complete clinical response refers to complete absence of the mass on physical exam, as well as absence of inflammation, ulceration and peau d'orange.

SECONDARY OUTCOMES:
Pathologic response | 6 months (approximately)
  Using the Residual Cancer Burden (RCB) index the pathologic response will be divided into categories. The three categories are complete response, near complete response and chemotherapy resistance. A complete pathologic response (pCR) refers to complete absence of invasive cancer.
Imaging Quantification | 6 months (approximately)
  Fluorothymidine Positron Emission Tomography (FLT PET) and Blood Oxygen Level Dependent (BOLD) MRI quantification of tumor responses to predict which patients are likely to achieve a pathologic complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Som Mukherjee, Principal Investigator — Juravinski Cancer Centre Hamilton, Ontario
Locations (4):
- Canada (4):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centres - London Regional Cancer Program, London, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Odette Health Sciences Centre, Toronto, Ontario